CLINICAL TRIAL: NCT00849381
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK580299) in Female Brazilian, Taiwanese and Thai Subjects Who Had Received Control Vaccine in Study 580299/008
Brief Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine in 580299/008 Subjects From Brazil, Taiwan or Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111758
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-08

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; HPV vaccine; papillomavirus; cervical cancer; human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

ARMS (2):
- Cervarix Compliance Issue Centre Group (Experimental): Subjects from one centre where compliance issues were discovered, who received the Hepatitis A control vaccine in the primary study (NCT00122681) and the Cervarix vaccine in the current study
  Interventions: Biological: GSK580299, GSK Biological's HPV vaccine
- Cervarix All Centres Group (Experimental): Subjects from all study centres who received the Hepatitis A control vaccine in the primary study (NCT00122681) and the Cervarix vaccine in the current study.
  Interventions: Biological: GSK580299, GSK Biological's HPV vaccine

INTERVENTIONS:
Biological: GSK580299, GSK Biological's HPV vaccine — All subjects will receive 3 doses administered as an intramuscular injection, according to a 0, 1, 6-month schedule.
  Other Names: CervarixTM

SUMMARY:
This phase 3b study is designed to assess the safety of GlaxoSmithKline Biological's HPV vaccine GSK580299 in female subjects who took part in study 008/580299 and received the control vaccine (Hepatitis A vaccine).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study
* A subject previously enrolled in the primary study (NCT00122681), who received the active control hepatitis A vaccine, and who cannot receive commercially available HPV-16/18 L1 VLP AS04 vaccine because the vaccine has not yet been granted licensure in the subject's country or because the subject is above the age for which the vaccine is licensed.
* Written informed consent must be obtained from the subject prior to enrolment.
* A woman aged 26 years or older at the time of the first vaccination in this study.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy should be verified with a urine pregnancy test.
* Subject must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or lactating female. Enrolment should be deferred until three months after pregnancy has been completed or after lactating has ceased.
* A woman planning to become pregnant or likely to become pregnant or planning to discontinue contraceptive prevention during the study period and up to two months after the last vaccine dose.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and the extended safety follow-up period.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product (pharmaceutical product or device).
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen by protocol.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days (i.e. Day 0-29) of each dose of vaccine. Administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous administration of components of the investigational vaccine.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex.
* Acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, haematological, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests, which in the opinion of the investigator precludes administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Cancer or autoimmune disease under treatment.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Acute disease at the time of enrolment.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1239 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Brazil (3):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Curitiba
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in this study were previously enrolled in the Control Group in the primary study (NCT00122681), where they had received Hepatitis A vaccination.
Pre-assignment Details: Results from one study center where compliance issues were discovered were presented both separately from the entire study cohort, as well as included in it. Out of the 1239 subjects enrolled in this study, 2 did not receive vaccination and were hence eliminated from the study.
Groups:
- Cervarix Group: Subjects who received the Hepatitis A control vaccine in the primary study (NCT00122681) and the Cervarix vaccine in the current study.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 1237 (Out of the subjects who started, 243 were enrolled at the center having compliance issues.)
Completed | 1092 (Out of the subjects who completed, 167 were enrolled at the center having compliance issues.)
Not Completed | 145
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 129
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 6
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 1237
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.2 (1.47)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Non-compliant center population
  Years | 28.7 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1237
  Male | 0
Gender [Number; unit: Participants] — Non-compliant center population
  Participants
    Female | 243
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
  Note: Results from one center where compliance issues were discovered are presented also separately.
Time Frame: During the entire study period (up to Month 12)
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 1237
Subjects
  Any SAEs all centers | 11
  Grade 3 SAEs all centers | 1
  Related SAEs all centers | 0
  Any SAEs non-compliant center (n=243) | 1
  Grade 3 SAEs non-compliant center (n=243) | 0
  Related SAEs non-compliant center (n=243) | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: MSCs include adverse events prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: During the entire study period (up to Month 12)
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 1237
Subjects
  Any MSCs all centers | 45
  Grade 3 MSCs all centers | 1
  Related MSCs all centers | 0
  Any MSCs non-compliant center (n=243) | 1
  Grade 3 MSCs non-compliant center (n=243) | 0
  Related MSCs non-compliant center (n=243) | 0

3. Primary Outcome: Number of Subjects With Pregnancies and Pregnancy Outcomes
Description: The pregnancy outcomes reported included elective termination, live birth and spontaneous abortion, all of which occurred with no apparent congenital (congenit.) anomalies (anom.) Note: Results from one non-compliant center (NCC) are also presented separately.
Time Frame: During the entire study period (up to Month 12)
Population: The analysis was based on the subjects with positive pregnancy results in the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of Cervarix vaccine in this study and for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 52
Subjects
  Elective termination NO congenit. anom. | 5
  Live infant NO apparent congenit. anom. | 40
  Lost to follow up | 2
  Spontaneous abortion NO congenit. anom. | 4
  Pregnancy Ongoing | 1
  Elective termination NO congenit. anom.(NCC, n=25) | 0
  Live infant NO apparent congenit. anom.(NCC, n=25) | 22
  Lost to follow up (NCC, n=25) | 1
  Spontaneous abortion NO congenit. anom.(NCC, n=25) | 1
  Pregnancy Ongoing (NCC, n=25) | 1

ADVERSE EVENTS:
Time Frame: SAEs were collected from study start until study end at Month 12.
Description: Other adverse events were not assessed in this study.
Arm/Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 11/1237
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=1237)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 3
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1
Appendicitis (Renal and urinary disorders) | 1
Chronic tonsillitis (Infections and infestations) | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombophlebitis (Vascular disorders) | 1
Thyroid cyst (Endocrine disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.